CLINICAL TRIAL: NCT04564989
Title: LCCC 2044: Prospective Observational Study to Validate Circulating HPVDNA and Prognostic Genomic Biomarkers in HPV-associated OPSCC
Brief Title: Prospective Observational Study to Validate Circulating HPVDNA and Prognostic Genomic Biomarkers in HPV-associated OPSCC
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Mayo Clinic (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 2044; 1U01DE029754-01 (NIH)
Record Dates: First submitted 2020-08-14; First posted 2020-09-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma; Carcinoma, Squamous Cell; Head and Neck Squamous Cell Carcinoma; Oropharynx Squamous Cell Carcinoma
Keywords: Human Papillomavirus; HPV; p16; Oropharynx; OPSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HPV+ OPSCC Patients: Patients with p16+ squamous cell carcinoma of the oropharynx (or unknown primary) who will receive definitive cancer treatment.

SUMMARY:
The primary goal of this study is to examine whether recurrence of HPV-associated OPSCC can be predicted by two factors: 1) mutations in genes called TRAF3 and CYLD, and 2) measurements of circulating HPV DNA in blood plasma. The study will also investigate whether HPV integration is associated with TRAF3 and CYLD mutations, and whether recurrence prediction improves when looking at HPV integration along with TRAF3 and CYLD mutations.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* T0-T2 N2a-N3 M0 or T3-T4 N0-N3 M0 (AJCC 7th edition)
* Biopsy proven squamous cell carcinoma of the oropharynx or unknown primary
* No prior therapy
* No evidence of distant metastatic disease
* p16 positive = diffuse ≥ 70% tumor cell expression, with at least moderate (2/3+) staining intensity
* Planned for receipt of definitive cancer treatment
* ECOG Performance Status 0-1
* Patients must be deemed able to comply with the treatment plan and follow-up schedule.
* Patients must provide study specific informed consent prior to study entry

Exclusion Criteria: All subjects meeting any of the exclusion criteria at baseline will be excluded from study participation:

* Prior history of radiation therapy to the head and neck
* Prior history of head and neck cancer.
* Inadequate pre-treatment tissue sample for tumor genomic analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HPV+ oropharyngeal squamous cell carcinoma who will receive definitive cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2033-11 (Estimated); Study Completion 2033-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence of OPSCC | From date of therapy completion until biopsy-proven recurrence, assessed up to 5 years
  Patients will undergo post-treatment CT scans per institutional standard of care to detect cancer recurrence. Status of recurrence of OPSCC will be confirmed based on biopsy.
Progression-free survival | From beginning or end of treatment until date of CT-detected recurrence or date of death, assessed up to 5 years
  Time-to-recurrence will be defined as time lapsed from end (or start) of treatment to first date recurrence (biopsy proven occur later) is detected by CT scans, or death. Otherwise, time-to-recurrence is censored at end of study date.
Positive Predictive Value | Baseline to up to 5 years
  Positive Predictive Value (PPV) is defined as probability that patients with two consecutive positive cHPVDNA (i.e., detectable cHPVDNA) really develop OPSCC recurrence during the study period.
Negative Predictive Value | Baseline to up to 5 years
  Negative Predictive Value (NPV) is defined as probability that patients without two consecutive positive cHPVDNA do not develop OPSCC recurrence during the study period.
Quality of Life questionnaire | Baseline until recurrence or up to 5 years
  At specified timepoints before, during, and after treatment, patients will complete a questionnaire comprised of questions from the European Organization for Research and Treatment of Cancer (EORTC) QLQ H&N35, which is for head and neck cancer patients, and EORTC QLQ C30, which is a general cancer assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Wendell Yarbrough, MD, Principal Investigator — UNC Chapel Hill
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Trident Medical Center (HCA Healthcare ), North Charleston, South Carolina

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials